CLINICAL TRIAL: NCT04333251
Title: Evaluating Convalescent Plasma to Decrease Coronavirus Associated Complications. A Phase I Study Comparing the Efficacy and Safety of High-titer Anti-Sars-CoV-2 Plasma vs Best Supportive Care in Hospitalized Patients With Interstitial Pneumonia Due to COVID-19
Brief Title: Study Testing Convalescent Plasma vs Best Supportive Care
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding was not obtained and study was not activated
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020-123
Record Dates: First submitted 2020-03-27; First posted 2020-04-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- convalescent plasma (Experimental): This arm will receive convalescent plasma
  Interventions: Biological: high-titer anti-Sars-CoV-2 plasma
- best supportive care (Placebo Comparator): Oxygen therapy
  Interventions: Other: oxygen therapy

INTERVENTIONS:
Biological: high-titer anti-Sars-CoV-2 plasma — Recipients will receive 1-2 units of ABO matched donor plasma at neutralization antibody titer >1:64 vs best supportive care
  Arms: convalescent plasma
Other: oxygen therapy — oxygen therapy
  Arms: best supportive care

SUMMARY:
Currently there are no proven treatment option for COVID-19. Human convalescent plasma is an option for COVID-19 treatment and could be available from people who have recovered and can donate plasma.

DETAILED DESCRIPTION:
Experience from prior outbreaks with other coronaviruses, such as SARS-CoV-1 shows that convalescent plasma contains neutralizing antibodies to the relevant virus. In the case of SARS-CoV-2, the anticipated mechanism of action by which passive antibody therapy would mediate protection is viral neutralization. The only antibody type that is currently available for immediate use is that found in human convalescent plasma. As more individuals contract COVID-19 and recover, the number of potential donors will continue to increase. The investigators seek to treat participants who are sick enough to warrant hospitalization prior to the onset of overwhelming disease.

ELIGIBILITY:
Inclusion Criteria Donor:

* 18 years or older
* must have been hospitalized w/COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing but are now PCR negative by 2 nasopharyngeal testing
* females of child-bearing potential must have a negative serum pregnancy test
* subject and/or LAR willing to provide informed consent
* patient agrees to storage of specimens for future testing

Inclusion Criteria Recipient:

* 18 years or older
* must have been hospitalized w/COVID-19 respiratory symptoms within 3 to 7 days from the beginning of illness
* subject and/or LAR willing to provide informed consent
* patient agrees to storage of specimens for future testing

Exclusion Criteria:

* 18 years or older
* receipt of pooled immunoglobulin in past 30 days
* contraindication to transfusion or history of prior reactions to transfusion blood products
* females who are identified as donors must not be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
reduction in oxygen and ventilation support | through study completion, an average of 4 weeks
  reduction in oxygen and ventilation support